CLINICAL TRIAL: NCT02227251
Title: A Phase 2b Open-label Study of Selinexor (KPT-330) in Patients With Relapsed/Refractory Diffuse Large B-Cell Lymphoma (DLBCL)
Brief Title: Selinexor (KPT-330) in Patients With Relapsed/Refractory Diffuse Large B-Cell Lymphoma (DLBCL)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCP-330-009; 2014-001977-15 (EudraCT Number)
Record Dates: First submitted 2014-08-12; First posted 2014-08-28 (Estimated); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: Diffuse large B-cell Lymphoma; DLBCL; Karyopharm; KPT-330; selinexor
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Part 1: Selinexor 60 mg (Experimental): Participants received fixed dose of 60 mg selinexor orally, twice weekly (BIW) on Days 1 and 3 (e.g., Monday and Wednesday or Tuesday and Thursday, etc.) of Weeks 1-4 of each four week (each cycle of 28 days) cycle (total of 8 doses per cycle).
  Interventions: Drug: Selinexor
- Part 2: Arm A-Selinexor 40 mg (Experimental): Participants received selinexor 40 mg orally BIW on Days 1 and 3 of each week of 4-week treatment cycles (28 days) until disease progression (total of 8 doses per cycle).
  Interventions: Drug: Selinexor
- Part 2: Arm B-Selinexor 60 mg (Experimental): Participants received selinexor 60 mg orally BIW on Days 1 and 3 of each week of 4-week treatment cycles) for 2 cycles (each cycle of 28 days) followed by 60 mg once weekly (QW) in the subsequent cycles until disease progression (total of 8 doses per cycle).
  Interventions: Drug: Selinexor

INTERVENTIONS:
Drug: Selinexor — Dose: 60 mg (BIW); Dosage form: film-coated (20 mg each) immediate release tablets; Route of administration: Oral
  Other Names: KPT-330
  Arms: Part 1: Selinexor 60 mg
Drug: Selinexor — Dose: 40 mg (BIW); Dosage form: film-coated (20 mg each) immediate release tablets; Route of administration: Oral
  Other Names: KPT-330
  Arms: Part 2: Arm A-Selinexor 40 mg
Drug: Selinexor — Dose: 60 mg (BIW) and 60 mg (QW); Dosage form: film-coated (20 mg each) immediate release tablets; Route of administration: Oral
  Other Names: KPT-330
  Arms: Part 2: Arm B-Selinexor 60 mg

SUMMARY:
A multicenter, open-label Phase 2b study of selinexor (KPT-330) in participants with relapsed/refractory (R/R) diffuse large B-cell lymphoma (DLBCL) who have no therapeutic options of demonstrated clinical benefit.

DETAILED DESCRIPTION:
This is a multicenter, open label, Phase 2b study of the selective inhibitor of nuclear export (SINE) selinexor (40 or 60 milligrams [mg]) given orally (PO) to participants with R/R DLBCL). The study is being conducted in 2 parts (Part 1 and Part 2). For Part 1, a fixed 60 mg dose of selinexor is given orally to 130 participants with R/R DLBCL who have no therapeutic options of demonstrated clinical benefit and who meet eligibility criteria and have none of the exclusion criteria will be enrolled to receive selinexor until either disease progression or intolerance has occurred. For Part 2, approximately 110 participants (55 in each arm) are planned to be enrolled. Participants will be randomized (open label) in a 1:1 ratio to either Arm A (40 mg) or Arm B (60 mg) and will be stratified based on history of prior autologous stem cell transplantation (ASCT) versus no prior ASCT. All the participants will be followed until disease progression and/or death.

ELIGIBILITY:
Inclusion Criteria (Parts 1 and 2):

* Written informed consent in accordance with federal, local, and institutional guidelines. The participant must provide informed consent prior to the first screening procedure.
* Age greater than or equal to (≥) 18 years.
* ECOG performance status of less than or equal to (≤) 2.
* Participants should have estimated life expectancy of greater than (>) 3 months at study entry.
* Previously treated, pathologically confirmed de novo DLBCL, or DLBCL transformed from previously diagnosed indolent lymphoma (e.g., follicular lymphoma).
* Participants must have received at least 2 but no more than 5 previous systemic regimens for the treatment of their de novo or transformed DLBCL including (i) at least 1 course of anthracycline-based chemotherapy (unless absolutely contraindicated due to cardiac dysfunction, in which case other active agents such as etoposide, bendamustine, or gemcitabine must have been given) and (ii) at least 1 course of anti-CD20 immunotherapy (e.g., rituximab), unless contraindicated due to severe toxicity. Participants who were considered ineligible for standard multi-agent immunochemotherapy must have received at least 2 and no more than 5 prior treatment regimens including at least 1 course of anti-CD20 antibodies and must be approved by the Medical Monitor. Prior stem cell transplantation is allowed; induction, consolidation, stem cell collection, preparative regimen and transplantation ± maintenance are considered a single line of therapy.
* Female participants of child-bearing potential must have a negative serum pregnancy test at screening and agree to use reliable methods of contraception for 3 months after their last dose of medication. Male participants must use a reliable method of contraception if sexually active with a female of child-bearing potential. For both male and female participants, effective methods of contraception must be used throughout the study and for 3 months following the last dose.

Part 1 additional inclusion criteria:

* For participants whose most recent systemic anti-DLBCL therapy induced a PR or CR, at least 60 days must have elapsed since the end of that therapy. For all other participants, at least 14 weeks (98 days) must have elapsed since the end of their most recent systemic anti-DLBCL therapy. . Palliative localized radiation within the therapy-free interval is allowed. Non-chemotherapy maintenance will not be considered anti DLBCL therapy, and therefore is allowed during the therapy-free interval.
* Documented clinical or radiographic evidence of progressive DLBCL prior to dosing.
* Participants must have measurable disease per the revised criteria for response assessment of lymphoma. Lymph nodes should be considered abnormal if the long axis is >1.5 centimeter (cm), regardless of the short axis. If a lymph node has a long axis of 1.1 to 1.5 cm, it should only be considered abnormal if its short axis is >1.0. Lymph nodes ≤1.0 by ≤1.0 will not be considered abnormal for relapse or PD.

Part 2 additional inclusion criteria:

• At least 3 weeks (21 days) must have elapsed since the end of participant's most recent systemic anti-DLBCL therapy (prior to Cycle 1 Day 1). Palliative localized radiation within the therapy-free interval is allowed.Non-chemotherapy maintenance will not be considered anti-DLBCL therapy, and therefore is allowed during the therapy-free interval.

• Adequate hematopoietic function: (i) Hemoglobin ≥10.0 grams per deciliters (g/dL) within 14 days of starting therapy (participant may receive red blood cell [RBC] transfusion within 14 days).

(ii) Absolute neutrophil count ≥1000 cells/millimeter (mm^3) (use of granulocyte growth factors prior to and during the study is acceptable).

(iii) Platelet count ≥100,000/mm^3 within 14 days of starting therapy (use of platelet growth factors prior to and during the study is acceptable).

* Participants must have measurable disease per the revised criteria for response assessment of lymphoma. Lymph nodes should be considered abnormal if the long axis is >1.5 cm, regardless of the short axis. Extranodal lesion should be considered abnormal if the long axis is >1.0 cm.

Exclusion Criteria (Parts 1 and 2):

* Participants who are pregnant or lactating.
* Primary mediastinal (thymic) large B-cell lymphoma (PMBL)
* Participants must not be eligible for high-dose chemotherapy with autologous stem cell transplantation rescue (Investigator must provide detailed documentation for ineligibility).
* Participants who have not recovered to Grade ≤1 clinically significant adverse events, or to their baseline, from their most recent systemic anti-DLBCL therapy.
* Major surgery within 2 weeks of first dose of study treatment.
* Participants with active hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV) infections.
* Psychiatric illness or substance use that would prevent the participant from giving informed consent or being compliant with the study procedures.
* Any of the following laboratory abnormalities:

  (i) A circulating lymphocyte count of >50,000/L. (ii) Hepatic dysfunction: bilirubin >2.0 times the upper limit of normal (ULN) (except participants with Gilbert's syndrome: total bilirubin of >3*ULN) and alanine aminotransferase (ALT) and aspartate aminotransferase (AST) >2.5 times ULN. In participants with known liver involvement of their DLBCL, AST and ALT >5*ULN.

(iii) Severe renal dysfunction: estimated creatinine clearance of <30 mL/min, measured in 24-hour urine or calculated using the formula of Cockroft and Gault [(140-Age)*Mass (kg)/(72*creatinine mg/dL); multiply by 0.85 if female].

* Any life-threatening illness, medical condition, or organ system dysfunction which, in the Investigator's opinion, could compromise the participant's safety.
* Participants with active graft-versus-host disease after allogeneic stem cell transplantation. At least 4 months must have elapsed since completion of allogeneic stem cell transplantation.
* Uncontrolled (i.e., clinically unstable) infection requiring parenteral antibiotics, antivirals, or antifungals on Cycle 1 Day 1; however, prophylactic use of these agents is acceptable even if parenteral.
* Participants unable to swallow tablets, participants with malabsorption syndrome, or any other gastrointestinal disease or gastrointestinal dysfunction that could interfere with absorption of study treatment.

Part 1 additional exclusion criteria:

* For participants whose most recent systemic anti-DLBCL therapy induced a PR or CR: Radiation, chemotherapy, immunotherapy, radio-immunotherapy, or any other anticancer therapy other than glucocorticoids <60 days or <14 weeks prior to Cycle 1 Day 1.
* Known central nervous system lymphoma or meningeal involvement.
* DLBCL with mucosa-associated lymphoid tissue [MALT] lymphoma, composite lymphoma (Hodgkin's lymphoma+NHL), or DLBCL transformed from diseases other than indolent NHL.
* Unstable cardiovascular function:

  (i) Symptomatic ischemia, or (ii) Uncontrolled clinically significant conduction abnormalities (i.e., ventricular tachycardia on anti-arrhythmia are excluded; 1st degree atrioventricular block or asymptomatic left anterior fascicular block /right bundle branch block will not be excluded), or (iii) Congestive heart failure of New York Heart Association Class ≥3, or (iv) Myocardial infarction within 3 months.
* Participants with a BSA <1.4 m^2 as calculated per Dubois 1916 or Mosteller 1987.
* Any of the following laboratory abnormalities:

  (i) Absolute neutrophil count (ANC) <1000 cells/mm^3 or platelet count <75,000/mm^3 during screening and on Cycle 1 Day 1. Use of granulocyte-stimulating factors and platelet growth factors prior to and during the study is acceptable.

(ii) Hematopoietic dysfunction: hemoglobin < 10.0 g/dL within 14 days of and including Cycle 1 Day 1 and/or patients receiving red blood cell (RBC) transfusion within 14 days of and including Cycle 1 Day 1.

* Participants who have been committed to an institution by official or judicial order.
* Participants with dependency on the Sponsor, Investigator or study site.

Part 2 additional exclusion criteria:

* Participants with active HBV, HVC, or HIV infections. Participants with active HBV are allowed if antiviral therapy for hepatitis B has been given for >8 weeks and viral load is <100 International units per milliliters (IU/mL) prior to first dose of study treatment. Participants with known history of HCV or found to be HCV antibody positive on screening, are allowed if there is documentation of negative viral load per institutional standard. Participants with HIV who have CD4+T-cell counts ≥350 cells/microliter (mcL), negative viral load per institutional standard, and no history of acquired immune deficiency syndrome (AIDS)-defining opportunistic infections in the last year are allowed.
* Known active central nervous system lymphoma or meningeal involvement. Participants with a history of CNS disease treated into remission may be enrolled.
* DLBCL with MALT lymphoma, composite lymphoma (Hodgkin's lymphoma + NHL), DLBCL arising from CLL (Richter's transformation), or high-grade B-cell lymphoma.
* Received strong cytochrome P450 3A (CYP3A) inhibitors ≤7 days prior to Day 1 dosing or strong CYP3A inducers ≤14 days prior to Day 1 dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2014-11 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Part 1: Overall Response Rate (ORR) | One year
  Assessed according to the revised response criteria based on the Guidelines of the International Working Group (IWG).
Part 2: Overall Response Rate (ORR) Based on Lugano Criteria | From initial randomization until date of disease progression or death (maximum of 1 year from Part 2 randomization)
  Assessed according to the response assessment of lymphoma based on Lugano classification.

SECONDARY OUTCOMES:
Part 1: Duration of Response (DOR) | From time of first response until disease progression or death (maximum of 1 year from Part 1 randomization)
Part 1: Disease Control Rate (DCR) | From initial response until disease progression or death (maximum of 1 year from Part 1 randomization)
Part 1: Number of Participants with Treatment-emergent Adverse Events (TEAEs) | From Baseline up to 30 days after last dose (maximum of 1 year from Part 1 randomization)
Part 1: Number of Participants with Eastern Cooperative Oncology Group (ECOG) Performance Status | From Baseline up to 30 days after last dose (maximum of 1 year from Part 1 randomization)
Part 2: Duration of response (DOR) | From time of first response (Part 2) until disease progression or death (maximum of 1 year from Part 2 randomization)
Part 2: Disease control rate (DCR) | From initial response (Part 2) until disease progression or death (maximum of 1 year from Part 2 randomization)
Part 2: Overall Response Rate (ORR) Based on Modified Lugano Criteria | From initial randomization until date of disease progression or death (maximum of 1 year from Part 2 randomization)
Part 2: Number of Participants with Treatment-emergent Adverse Events | From Baseline up to 30 days after last dose (maximum of 1 year from Part 2 randomization)
Part 2: Number of Participants with Eastern Cooperative Oncology Group (ECOG) Performance Status | From Baseline up to 30 days after last dose (maximum of 1 year from Part 2 randomization)

CONTACTS AND LOCATIONS:
Locations (176):
- United States (23):
  - UACC Arizona, Tucson, Arizona
  - University of California San Francisco, San Francisco, California
  - University of California Los Angeles (UCLA), Santa Monica, California
  - Boca Raton Cancer Research Medical Center, Plantation, Florida
  - University of Chicago, Chicago, Illinois
  - Robert H. Lurie Comprehensive Cancer Center/Northwestern University, Chicago, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Clinical Research Alliance, Lake Success, New York
  - New York Presbyterian Hospital/ Cornell Medical College, New York, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Gabrail Cancer Center, Canton, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University Hospitals Seidman Cancer Center, Cleveland, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Greenville Hospital System, Greenville, South Carolina
  - MD Anderson, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington
  - Virginia Mason Hospital & Medical Center, Seattle, Washington
- Australia (11):
  - St. Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Liverpool Hospital, Ingham Institute of Medical Research, Liverpool, New South Wales
  - Calvary Mater Newcastle Hospital, Waratah, New South Wales
  - Icon Cancer Care, South Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Ashford Cancer Centre, Kurralta Park, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - Epworth Hospital, East Melbourne, Victoria
  - St. Vincent's Melbourne, Fitzroy, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Austria (9):
  - Medical University of Graz, Graz
  - Medizinische Universität Innsbruck für Innere Medizin, Innsbruck
  - LKH Leoben Department for Haemato-Oncology, Leoben
  - Akh Linz Innere Med III - Zentrum für Hämatologie und med. Onkologie, Linz
  - Krankenhaus Barmherzigen Schwestern Linz, Linz
  - Krankenhaus der Elisabethinen Linz GmbH, Linz
  - Uni. Klinik für Innere Medizin III Universitätsklinikum der PMU LKH Salzburg, Salzburg
  - Medical University of Vienna (MUW) Department of Medicine I, Vienna
  - Univ. General Hospital Hietzing, Vienna
- Belgium (8):
  - Ziekenhuis Netwerk Antwerpen, Antwerp
  - AZ Sint-Jan, Bruges
  - Institut Jules Bordet, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Gent, Ghent
  - CH Jolimont, La Louvière
  - AZ Delta, Roeselare
  - H-Hartziekenhuis Roeselare-Menen, Roeselare
- Bulgaria (3):
  - University Hospital for Active Treatment Dr. Georgi Stranski, Pleven
  - University Multiprofile Hospital for Active Treatment Sveti Ivan Rilski EAD, Sofia
  - Specialized Hospital for Active Treatment of Haematological Diseases EAD, Sofia
- Canada (2):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Sir Mortimer B Davis Jewish General Hospital/McGill University, Montreal, Quebec
- France (12):
  - CHU Lyon Sud, Pierre-Bénite, Lyon
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - Unite Hemopathies Lymphoides Chu Henri Mondor, Créteil
  - Chu Dijon-Bourgogne - Hematologie Clinique, Dijon
  - Hospitalier de la Rochelle-Ré-Aunis, La Rochelle
  - CHRU de Lille - Hopital Claude-Huriez, Lille
  - Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille
  - CHU Montpellier, Montpellier
  - Hostpial Saint Louis - CIRCO (Centre d'Investigations et de Recherche Clinique en Oncologie), Paris
  - Hôpital Necker Service d'Hématologie Adult, Paris
  - Pitié-Salpêtrière Hospital, Paris
  - Centre Henri Becquerel, Rouen
- Germany (14):
  - Uniklinik Aachen Klinik für Hämatologie, Onkologie, Hämostaseologie und Stammzelltransplantation, Aachen
  - HELIOS Klinikum Bad Saarow, Bad Saarow
  - Charite Universitatsmedizin Berlin (Benjamin Franklin Campus), Berlin
  - Charite Universitatsmedizin Berlin (Virchow Campus), Berlin
  - Ev. Diakonie-Krankenhaus gGmbH, Bremen
  - Klinikum Kempten Klinik für Innere Medizin III - Hämatologie, Onkologie und Palliativmedizin, Cologne
  - Gemeinschaftspraxis Haematologie and Onkologie-Dresden, Dresden
  - Martin-Luther-University Halle-Wittenberg Department of Oncology, Halle
  - Medizinische Hochschule, Hanover
  - Universität Heidelberg Medizinische Klinik V Hämatologie, Onkologie und Rheumatologie, Heidelberg
  - Klinikum Leverkusen, Leverkusen
  - Klinikum Ludwigshafen, Ludwigshafen
  - Rotkreuzklinikum München, München
  - Klinikum Nürnberg Nord, Nuremberg
- Greece (8):
  - Haematology Department and HCT Unit G.Papanicolaou Hospital, Exochi, Thessaloniki
  - Hematology Clinic,General Hospital of Athens,G. Gennimatos, Athens
  - National & Kapodistrian University of Athens, Laiko General Hospital, Athens
  - Hematology Department Laiko General Hospital, Athens
  - Second Depth of Internal Medicine, Attiko University Hospital, Athens
  - National & Kapodistrian University of Athens, Attiko University Hospital, Chaïdári
  - Department of clinical hematology ,university hospital Ioannina, Ioannina
  - University of Patras Medical School, Pátrai
- Hungary (7):
  - Semmelweis Egyetem Általános Orvosi Kar, Budapest
  - Országos Onkológiai Intézet "A" Belgyógyászati Onkológiai Osztály, Budapest
  - Semmelweis University Department of Medicine and Oncology, Budapest
  - Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár
  - Pécsi Tudományegyetem, ÁOK, I. számú Belgyógyászati Klinika, Pécs
  - Veszprém Megyei Csolnoky Ferenc Kórház, Veszprém
  - CSolnoky ferenc Hospital, Veszprém
- India (20):
  - Regional Cancer Centre, IGIMS, Patna, Bihar
  - SRM Institutes for Medical Science, Vadapalani, Chennai
  - IRCH, All India Institute of Medical Sciences, Delhi, India
  - Regional Cancer Centre, Thiruvananthapuram, Kerala
  - Prince Aly Khan Hospital, Mumbai, Maharashtra
  - Jaslok Hospital and Research Centre, Mumbai, Maharashtra
  - Deenanath Mangeshkar Hospital, Pune, Maharashtra
  - Rajiv Gandhi Cancer Hospital, New Delhi, National Capital Territory of Delhi
  - Institute of Medical Sciences & SUM Hospital, Bhubaneswar, Odisha
  - Dayanand Medical College and Hospital, Ludhiana, Punjab
  - Cancer Institute (WIA), Chennai, Tamil Nadu
  - Saveetha Medical College Hospital, Chennai, Tamil Nadu
  - G. Kuppu Swamy Naidu Hospital, Coimbatore, Tamil Nadu
  - Meenakshi Mission Hospital & Research Centre, Madurai, Tamil Nadu
  - King George's Medical University (KGMU), Lucknow, Uttar Pradesh
  - Nil Ratan Sircar Medical College and Hospital, Kolkata, West Bengal
  - Netaji Subhas Chandra Bose Cancer Research Hospital, Kolkata, West Bengal
  - TATA Memorial Centre, Kolkata, West Bengal
  - Netaji Subhas Chandra Bose Cancer Research Institute, Kolkata, West Bengal
  - Dr. B.R.A. Institute Rotary Cancer Hospital All India Institute of Medical Sciences, New Delhi
- Israel (8):
  - Hematology-Soroka, Beersheba
  - Rambam Healthcare Campus, Haifa
  - Wolfson MC, Holon
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Assuta Medical Center, Tel Aviv
  - TLV Sorasky Medical Center, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky
- Italy (8):
  - Instituto di Ematologia Seragnoli Pad 8 Universita di Bologna, Bologna
  - SODc Ematologica ,AOU Careggi, Florence
  - AOU Maggiore della Carità SCDU Ematologia, Florence
  - Hematology-Oncology & Stem Cell Transplantation Unit, National Cancer Institute, Fondazione 'G. Pascale', IRCCS, Naples
  - SCDU Ematologia, Division of Hematology, Dept. of Translational Medicine, Universita del Piemonte Orientale, Novara
  - Fondazione Policlinico Universitario A. Gemelli, Rome
  - Azienda Ospedaliero-Universitaria Senese, Siena
  - Città della Salute e della Scienza di Torino, Torino
- Netherlands (2):
  - VUMc (Vrije Universiteit Amsterdam), Amsterdam
  - LUMC (leidse universitair medisch centrum), Leiden
- New Zealand (2):
  - North Shore Hospital, Auckland
  - Christchurch Hospital, Christchurch
- Poland (11):
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza, Wroclaw, Radeckiego
  - Szpitale Wojewódzkie w Gdyni, Gdyńskie Centrum onkologii, Gdynia
  - MCM (Małopolskie Centrum Medyczne), Krakow
  - Wojewodzki Szpital Specjalistyczny w Legnicy, Legnica
  - Memorial Provincial Specialist Hospital in Lodz, Lodz
  - Samodzielny Publiczny Szpital Kliniczny nr 1 w Lublinie, Lublin
  - Hematology Department St John's Cancer Centre, Lublin
  - Samodzielny Publiczny Zakład Opieki Zdrowotnej Ministerstwa, Olsztyn
  - Instytut Hematologii i Transfuzjologii, Warsaw
  - Centrum Onkologii- Insytut Im. Marii Skłodowskiej-Curie Klinika Nowotworow Ukladu Chlonnego, Warsaw
  - Maria Sklodowska Curie National Research Institute, Warsaw
- Serbia (6):
  - Institut za onkologiju i radiologiju Srbije, Belgrade
  - Klinicko Bolnick Centar Zemun Odeljenje hematologije, Belgrade
  - Klinički centar Srbije Klinika za hematologiju, Belgrade
  - Kliničko bolnički centar Zvezdara, Belgrade
  - Institut za onkologiju Vojvodine, Kamenitz
  - Klinički centar Niš Klinika za hematologiju, Niš
- Spain (8):
  - Hospitla Universitari Germans Trias i Pujol - ICO, Badalona
  - Hospital University Vall d'Hebron, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital de Son Llàtzer, Palma de Mallorca
  - Clínica Universidad De Navarra, Pamplona
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocio, Seville
- United Kingdom (14):
  - Gloucestershire Royal Hospital, Gloucester, Gloucestershire
  - Southampton University Hospital, Southampton, Hampshire
  - Royal Marsden Hospital, Sutton, London
  - Northwick Park Hospital, Harrow, Middlesex
  - Leeds Teaching Hospitals NHS Trust, Leeds, Yorkshire
  - Addenbrooke's Hospital Cambridge, Cambridge
  - Royal Liverpool University Hospital, Liverpool
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool
  - King's College Hospital, London
  - Princess Royal University Hospital (PRUH), London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - Oxford University Hospitals NHS Trust Oxford Cancer and Haematology Centre, Churchill Hospital, Oxford
  - Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schuster M, Zijlstra J, Casasnovas RO, Vermaat JSP, Kalakonda N, Goy A, Choquet S, Neste EVD, Hill B, Thieblemont C, Cavallo F, De la Cruz F, Kuruvilla J, Hamad N, Jaeger U, Caimi P, Gurion R, Warzocha K, Bakhshi S, Sancho JM, Follows G, Egyed M, Offner F, Vassilakopoulos T, Samal P, Ku M, Ma X, Corona K, Chamoun K, Shah J, Shacham S, Kauffman MG, Canales M, Maerevoet M. Effect of Prior Therapy and Disease Refractoriness on the Efficacy and Safety of Oral Selinexor in Patients with Diffuse Large B-cell Lymphoma (DLBCL): A Post-hoc Analysis of the SADAL Study. Clin Lymphoma Myeloma Leuk. 2022 Jul;22(7):483-494. doi: 10.1016/j.clml.2021.12.016. Epub 2021 Dec 25. PMID 35078739
- [Derived] Maerevoet M, Zijlstra JM, Follows G, Casasnovas RO, Vermaat JSP, Kalakonda N, Goy A, Choquet S, Van Den Neste E, Hill B, Thieblemont C, Cavallo F, De la Cruz F, Kuruvilla J, Hamad N, Jaeger U, Caimi P, Gurion R, Warzocha K, Bakhshi S, Sancho JM, Schuster M, Egyed M, Offner F, Vassilakopoulos TP, Samal P, Ku M, Ma X, Corona K, Chamoun K, Shah J, Shacham S, Kauffman MG, Canales M. Survival among patients with relapsed/refractory diffuse large B cell lymphoma treated with single-agent selinexor in the SADAL study. J Hematol Oncol. 2021 Jul 16;14(1):111. doi: 10.1186/s13045-021-01122-1. PMID 34271963
- [Derived] Shah J, Shacham S, Kauffman M, Daniele P, Tomaras D, Tremblay G, Casasnovas RO, Maerevoet M, Zijlstra J, Follows G, P Vermaat JS, Kalakonda N, Goy AH, Choquet S, Den Neste EV, Hill BT, Thieblemont C, Cavallo F, la Cruz F, Kuruvilla J, Hamad N, Bouabdallah R, Jager U, Caimi P, Gurion R, Warzocha K, Bakhshi S, Sancho JM, Schuster M, Egyed M, Offner F, Vasilakopoulos TP, Samal P, Nagy A, Ku M, Canales Albendea MA. Health-related quality of life and utility outcomes with selinexor in relapsed/refractory diffuse large B-cell lymphoma. Future Oncol. 2021 Apr;17(11):1295-1310. doi: 10.2217/fon-2020-0946. Epub 2021 Feb 2. PMID 33528286
- [Derived] Kalakonda N, Maerevoet M, Cavallo F, Follows G, Goy A, Vermaat JSP, Casasnovas O, Hamad N, Zijlstra JM, Bakhshi S, Bouabdallah R, Choquet S, Gurion R, Hill B, Jaeger U, Sancho JM, Schuster M, Thieblemont C, De la Cruz F, Egyed M, Mishra S, Offner F, Vassilakopoulos TP, Warzocha K, McCarthy D, Ma X, Corona K, Saint-Martin JR, Chang H, Landesman Y, Joshi A, Wang H, Shah J, Shacham S, Kauffman M, Van Den Neste E, Canales MA. Selinexor in patients with relapsed or refractory diffuse large B-cell lymphoma (SADAL): a single-arm, multinational, multicentre, open-label, phase 2 trial. Lancet Haematol. 2020 Jul;7(7):e511-e522. doi: 10.1016/S2352-3026(20)30120-4. PMID 32589977